CLINICAL TRIAL: NCT01970657
Title: An Observational Study Providing 12 Months of Safety Follow-Up From First Exposure to HP802-247 in Subjects Who Participated in Study 802-247-09-032(EU)
Brief Title: Observational Study Providing 12 Months of Safety Follow-Up From First Exposure to HP802-247
Status: Completed | Type: Observational
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Other Study IDs: 802-247-09-033
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Venous Leg Ulcer (VLU)
Keywords: Venous Stasis Ulcer; VLU
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — The treatment assignment codes and randomization schedule for the prior trial will be maintained for this observational study. The treatment assignments will not be made known to the Investigators until the present follow-up study has been completed by all consenting subjects thus keeping treating physician and subjects blind to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HP802-247 in prior study: Observational safety follow up study, no treatment specified
  Interventions: Biological: No treatment specified
- Vehicle Control in prior study: Observational safety follow up study, no treatment specified
  Interventions: Biological: No treatment

INTERVENTIONS:
Biological: No treatment specified — No intervention
  Groups: HP802-247 in prior study
Biological: No treatment — None specified
  Groups: Vehicle Control in prior study

SUMMARY:
This observational safety follow-up study enrolled subjects from the 802-247-09-032 study with the investigational product HP802-247 for venous leg ulcers, who received at least one application of HP802-247 or Vehicle (Placebo). This study is being done for the following purposes:

1. to identify new adverse events,
2. to examine ongoing adverse events not resolved in subjects who participated in the 802-247-09-032 trial,
3. to record wound status, and
4. to determine if there are differences in Health Related Quality of Life (HRQoL) associated with the treatment assignment from the 802-247-09-032 Trial.

About 440 subjects were to participate depending upon subject enrollment from the previous study, 802-247-09-032. The study was conducted in approximately 50 sites in Europe.

DETAILED DESCRIPTION:
Subjects transitioned to this observational study immediately upon exit from the 802-247-09-032 trial. This ensured a total of 12 months of safety observations and wound status data were obtained from the time of the first application of HP802-247. This study provided consecutive visits at intervals of 8 weeks until a total of 12 months of safety follow-up had been achieved, based on the initial application of Investigational Medicinal Product in the prior study. Specifically, this study examines all new and unresolved ongoing adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent document must be read, signed, and dated by the subject or the subject's legally authorized representative before conducting any study procedures or exams.
* Subject was randomized in 802-247-09-032 and received at least one application of test article.
* Subject has ended their participation in 802-247-09-032 by virtue of completing the study, or by dropping out prior to completion.

Exclusion Criteria:

* Subjects who refuse to provide written informed consent for this study will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Assess new adverse events, and ongoing adverse events not resolved, in subjects who were exposed to a Investigational Medicinal Product in the 802-247-09-032 trial. | Up to 12 months from first application of test article in the 802-247-09-032 study
  The evaluation of safety included analysis of new test article-related events, as well as continued follow-up of those adverse events that originated in the prior study.

SECONDARY OUTCOMES:
Follow-up on the status of the target ulcer as open, re-opened or closed. | Up to 12 months from first application of test article in the 802-247-09-032 study
  At each study visit the status of the target ulcer was assessed as remaining closed, re-opened, or a new closure.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Vanscheidt, MD, Principal Investigator — University Freiburg-Practice for Dermatology
Locations (43):
- Belgium (3):
  - Brussels
  - Edegem
  - Ghent
- Czechia (9):
  - Brno
  - Hradec Králové
  - Olomouc
  - Pardubice
  - Plzen-Bory
  - Prague
  - Třebíč
  - Uherské Hradiště
  - Ústí nad Labem
- Germany (15):
  - Bochum
  - Bonn
  - Cologne
  - Dresden
  - Düsseldorf
  - Essen
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Hamburg
  - Kiel
  - Krefeld
  - Magdeburg
  - München
  - Münster
- Hungary (7):
  - Budapest
  - Debrecen
  - Hatvan
  - Orosháza
  - Sátoraljaújhely
  - Szeged
  - Szolnok
- Poland (9):
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Rzeszów
  - Studzionka
  - Warsaw
  - Wroclaw
  - Zabrze

IPD SHARING:
Plan to Share IPD: Yes
Publication submitted to Journal of Vascular Surgery in May 2017